CLINICAL TRIAL: NCT06956170
Title: A Phase III, Multicenter, Open-Label, Randomized Study to Evaluate the Efficacy and Safety of Belantamab Mafodotin in Combination With Pomalidomide and Dexamethasone (B-Pd) Versus Pomalidomide Plus Bortezomib and Dexamethasone (PVd) in Participants With Relapsed/Refractory Multiple Myeloma (DREAMM 8)
Brief Title: All Japanese Population: Belantamab Mafodotin Plus Pomalidomide and Dexamethasone (Pd) Versus Bortezomib Plus Pd in Relapsed/Refractory Multiple Myeloma
Acronym: DREAMM 8
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 207499-JPN
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Multiple Myeloma
Keywords: Japan population; Belantamab Mafodotin; Relapsed/Refractory Multiple Myeloma; Pomalidomide; Dexamethasone; Bortezomib
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; pomalidomide; Dexamethasone; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Belantamab mafodotin plus Pomalidomide and Dexamethasone (Experimental)
  Interventions: Drug: Belantamab mafodotin; Drug: Pomalidomide; Drug: Dexamethasone
- Bortezomib plus Pomalidomide and Dexamethasone (Active Comparator)
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone; Drug: Bortezomib

INTERVENTIONS:
Drug: Belantamab mafodotin — Humanized anti-B-cell maturation antigen (BCMA) antibody/drug conjugate will be administered.
  Arms: Belantamab mafodotin plus Pomalidomide and Dexamethasone
Drug: Pomalidomide — Immunomodulatory drug (IMiD) will be administered.
Drug: Dexamethasone — Synthetic glucocorticoid with anti-tumor activity will be administered.
Drug: Bortezomib — Proteasome Inhibitor will be administered.
  Arms: Bortezomib plus Pomalidomide and Dexamethasone

SUMMARY:
This study will evaluate the efficacy and safety of belantamab mafodotin in combination with pomalidomide and dexamethasone compared with that of combination of pomalidomide, bortezomib and dexamethasone in Japanese participants with relapsed/refractory multiple myeloma (RRMM).

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent.
* Male or female, 18 years or older.
* Have a confirmed diagnosis of multiple myeloma (MM) as defined by the International Myeloma Working Group (IMWG) criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Have been previously treated with at least 1 prior line of MM therapy including a lenalidomide-containing regimen and must have documented disease progression during or after their most recent therapy. (Participants treated with lenalidomide ≥10 mg daily for at least 2 consecutive cycles are eligible).
* Must have at least 1 aspect of measurable disease defined as one of the following;

  1. Urine M-protein excretion greater than or equal to (≥)200 milligrams (mg) per 24-hour, or
  2. Serum M-protein concentration ≥0.5 grams/deciliters (g/dL) (≥5.0 g/liter [L]), or
  3. Serum free light chain (FLC) assay: involved FLC level ≥10 mg/dL (≥100 mg/L) and an abnormal serum free light chain ratio (less than [<]0.26 or greater than [>]1.65) only if participant has no measurable urine or serum M spike.
* Have undergone autologous stem cell transplant (ASCT) or are considered transplant ineligible. Participants with a history of ASCT are eligible for study participation provided the following eligibility criteria are met: a. ASCT was >100 days prior to the first dose of study medication. b. No active bacterial, viral, or fungal infection(s) present
* All prior treatment-related toxicities (defined by National Cancer Institute Common Terminology Criteria for Adverse Events [NCI-CTCAE] version 5.0) must be less than or equal to (≤)Grade 1 at the time of enrolment, except for alopecia.
* Adequate organ system functions as mentioned in the protocol.
* Male and female participants agree to abide by protocol-defined contraceptive requirements.
* In Japan, Hepatitis B participants who are hepatitis B surface antigen (HbsAg)- (e.g. HBsAb+/HbsAg-, HBcAb+/HbsAg-, HBcAb+/HBsAb+/HbsAg-) are eligible for inclusion in this study if hepatitis B virus (HBV) DNA is undetectable. A patient with HBsAg+ is eligible if HBV DNA is undetectable after assessing hepatitis B e antigen (HBeAg), hepatitis B e antibody (HBeAb) and HBV DNA, and if a hepatologist agrees with the participation into this study.

Exclusion Criteria:

* Active plasma cell leukemia, symptomatic amyloidosis or active polyneuropathy, organomegaly, endocrinopathy, monoclonal plasma proliferative disorder, and skin changes (POEMS) syndrome at the time of screening.
* Prior allogeneic SCT.
* Systemic anti-myeloma therapy (including chemotherapy and systemic steroids) within 14 days or five half-lives (whichever is shorter) preceding the first dose of study drug; prior treatment with a monoclonal antibody drug within 30 days of receiving the first dose of study drugs.
* Plasmapheresis within 7 days prior to the first dose of study drug.
* Received prior treatment with or intolerant to pomalidomide.
* Received prior Beta cell maturation antigen (BCMA) targeted therapy.
* Intolerant to bortezomib or refractory to bortezomib (for example; participant experienced progressive disease during treatment, or within 60 days of completing treatment, with a bortezomib-containing regimen of 1.3 mg/meter square [m^2] twice weekly).
* Evidence of cardiovascular risk including any of the following;

  1. Evidence of current clinically significant untreated arrhythmias, including clinically significant electrocardiogram abnormalities including second degree (Mobitz type II) or third degree atrioventricular (AV) block.
  2. Recent history within (3 months of screening) of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting .
  3. Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system
  4. Uncontrolled hypertension.
* Any major surgery within the last 4 weeks.
* Previous or concurrent invasive malignancy other than multiple myeloma, except:

  1. The disease must be considered medically stable for at least 2 years; or
  2. The participant must not be receiving active therapy, other than hormonal therapy for this disease.
* Known immediate or delayed hypersensitivity reaction or idiosyncratic reaction to belantamab mafodotin or drugs chemically related to belantamab mafodotin, or any of the components of the study treatment.
* Evidence of active mucosal or internal bleeding.
* Cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice.
* Active infection requiring treatment.
* Known or active human immunodeficiency virus (HIV) infection, hepatitis B or hepatitis C will be excluded unless the protocol-defined criteria are met.
* Presence of active renal conditions (such as infection, severe renal impairment requiring dialysis or any other condition that could affect participant's safety).
* Ongoing Grade 2 peripheral neuropathy with pain within 14 days prior to randomization or ≥Grade 3 peripheral neuropathy.
* Active or history of venous and arterial thromboembolism within the past 3 months.
* Contraindications to or unwilling to undergo protocol-required anti-thrombotic prophylaxis.
* Current corneal disease except for mild punctate keratopathy.
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions (including laboratory abnormalities) that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures.
* Pregnant or lactating female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2029-11-30 (Estimated)

CONTACTS AND LOCATIONS:
Locations (13):
- Japan (13):
  - GSK Investigational Site, Nagoya, Aichi-ken
  - GSK Investigational Site, Kamogawa, Chiba
  - GSK Investigational Site, Kashiwa, Chiba
  - GSK Investigational Site, Matsuyama, Ehime
  - GSK Investigation Site, Fukushima, Fukushima
  - GSK Investigational Site, Maebashi, Gunma
  - GSK Investigational Site, Shibukawa, Gunma
  - GSK Investigational Site, Numakunai, Iwate
  - GSK Investigational Site, Okayama, Okayama-ken
  - GSK Investigational Site, Osaka, Osaka
  - GSK Investigational Site, Tottori-shi, Tottori
  - GSK Investigational Site, Yamagata, Yamagata
  - GSK Investigational Site, Hokkaido

IPD SHARING:
Plan to Share IPD: No
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled a total of 12 Japanese participants and the analyses included 9 Japanese participants that had been previously enrolled in the global study for 207499 (NCT04484623), resulting in a total of 21 participants.
Pre-assignment Details: The results presented are until the primary completion date. Additional results will be provided within a year of study completion.
Groups:
- Belantamab Mafodotin+Pomalidomide+Dexamethasone: Japanese participants with Relapsed/Refractory Multiple Myeloma (RRMM) received intravenous (IV) infusion of 2.5 milligram (mg)/kilogram (kg) belantamab mafodotin on Day 1 of Cycle 1 and 1.9 mg/kg on Day 1 of Cycle 2 onwards in each 28-day cycle, in combination with oral 4 mg per day Pomalidomide capsule on Days 1 to 21 of each 28-day cycle; and oral 40 mg per day Dexamethasone tablet on Days 1, 8, 15, and 22 of each 28-day cycle until disease progression, death, unacceptable toxicity, withdrawal of consent, initiation of another anti-myeloma therapy or end of study, whichever occurs first.
- Bortezomib + Pomalidomide + Dexamethasone: Japanese participants with RRMM received subcutaneous (SC) injection of 1.3 mg/meter^2(m^2) Bortezomib on Days 1, 4, 8, 11, of each 21-day cycle for Cycles 1 through 8, and on Days 1, 8, of each 21-day cycle for Cycles 9+ in combination with oral 4 mg per day Pomalidomide capsule on Days 1 to 14 of each 21-day cycle, and oral 20 mg Dexamethasone tablet on Days 1, 2, 4, 5, 8, 9, 11, 12, of each 21-day cycle for Cycles 1 through 8 and then on Days 1, 2, 8, 9, every 3 Weeks (Q3W) from Cycles 9 onwards until disease progression, death, unacceptable toxicity, withdrawal of consent, initiation of another anti-myeloma therapy or end of study, whichever occurs first.
Period: Overall Study
Arm/Group | Belantamab Mafodotin+Pomalidomide+Dexamethasone | Bortezomib + Pomalidomide + Dexamethasone
Started | 10 | 11
Completed | 0 | 0
Not Completed | 10 | 11
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Ongoing | 7 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Belantamab Mafodotin+Pomalidomide+Dexamethasone | Bortezomib + Pomalidomide + Dexamethasone | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 72.6 (5.95) | 72.5 (5.70) | 72.6 (5.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 4 | 5 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian- Japanese Heritage | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as time from randomization until earliest date of disease progression (PD), determined by Independent Review Committee (IRC), according to the International Myeloma Working Group (IMWG) Response Criteria, or death due to any cause. PD is defined as increase of >=25% from lowest value in >=1 of following (serum M-protein [absolute increase >=0.5 grams per deciliter {g/dL}]; serum M-protein increase >=1g/dL [when lowest M-protein >=5g/dL]; urine M-protein [absolute increase >=200 milligrams per 24 hours {mg/24h}]; participants without measurable serum & urine M-protein levels, difference between involved & uninvolved serum free light chains (sFLC) levels [absolute increase >10mg/dL]; appearance of new lesion,>=50% increase from nadir in Sum of the products of the maximal perpendicular diameters of measured lesions (SPD) of >1 lesion, or >=50% increase in longest diameter of previous lesion >1 centimeter (cm) in short axis.
Time Frame: Up to approximately 120 weeks
Population: Intent-to-Treat (ITT) Population included all randomized participants whether or not randomized treatment was administered.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Belantamab Mafodotin+Pomalidomide+Dexamethasone | Bortezomib + Pomalidomide + Dexamethasone
Number analyzed (Participants) | 10 | 11
Months | NA [0.2 to NA] — The median and upper limit of 95% Confidence Interval were not estimable due to an insufficient number of participants with events within the length of follow-up in assessing the number of events. | 14.8 [1.9 to NA] — The upper limit of 95% Confidence Interval was not estimable due to an insufficient number of participants with events within the length of follow-up in assessing the number of events.
Statistical Analysis 1: Comparison: Belantamab Mafodotin+Pomalidomide+Dexamethasone vs Bortezomib + Pomalidomide + Dexamethasone; Test type: Other; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.10 to 2.78] — Hazard ratio was estimated using an unstratified Cox Proportional Hazard model with treatment arm as an explanatory variable

2. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) defined as the interval of time from randomization to the date of death due to any cause.
Time Frame: Up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

3. Secondary Outcome: Duration of Response (DoR)
Description: Duration of Response (DoR) defined as the time from first documented evidence of partial response (PR) or better until progressive disease (PD) or death due to any cause. Response will be based on IRC-assessment per IMWG criteria.
Time Frame: Up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

4. Secondary Outcome: Minimal Residual Disease (MRD) Negativity Rate
Description: MRD negativity rate defined as the percentage of participants who achieve MRD negative status (as assessed by NGS at 10^5 threshold) at least once during the time of confirmed CR or better response based on IRC-assessment per IMWG.
Time Frame: Up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

5. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a confirmed partial response or better (i.e., PR, VGPR, CR, and sCR) based on IRC-assessment per IMWG criteria.
Time Frame: Up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

6. Secondary Outcome: Complete Response Rate (CRR)
Description: Complete Response Rate (CRR), defined as the percentage of participants with a confirmed complete response (CR) or better (i.e., CR and stringent complete response (sCR)) based on IRC assessment per IMWG criteria.
Time Frame: Up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

7. Secondary Outcome: Percentage of Participants With a Confirmed Very Good Partial Response (VGPR) or Better
Description: VGPR is defined as the percentage of participants with a confirmed VGPR or better (i.e., VGPR, CR, and sCR) based on IRC-assessment per IMWG criteria.
Time Frame: Up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

8. Secondary Outcome: Time to Best Response (TTBR)
Description: Time to Best Response (TTBR) defined as the interval of time between the date of randomization and the earliest date of achieving best response among participants with a confirmed PR or better based on IRC-assessment per IMWG.
Time Frame: Up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

9. Secondary Outcome: Time to Response (TTR)
Description: Time to Response (TTR) defined as the time between the date of randomization and the first documented evidence of response (PR or better) among participants who achieve a response (i.e., confirmed PR or better) based on IRC-assessment per IMWG.
Time Frame: Up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

10. Secondary Outcome: Time to Progression (TTP)
Description: Time to Progression (TTP) defined as the time from randomization until the earliest date of PD based on IRC-assessment per IMWG criteria, or death due to PD.
Time Frame: Up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

11. Secondary Outcome: Progression-free Survival on Subsequent Line of Therapy (PFS2)
Description: PFS2 defined as time from randomization to disease progression (investigator-assessed response) after initiation of new anti-myeloma therapy or death from any cause, whichever is earlier. If disease progression after new antimyeloma therapy cannot be measured, a PFS event is defined as the date of discontinuation of new anti-myeloma therapy, or death from any cause, whichever is earlier.
Time Frame: Up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

12. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA dictionary).
Time Frame: Up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

13. Secondary Outcome: Number of Participants With Clinically Significant Changes in Hematology Parameters
Description: Blood samples will be collected for the analysis of hematology parameters.
Time Frame: Up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

14. Secondary Outcome: Number of Participants With Clinically Significant Changes in Clinical Chemistry Parameters
Description: Blood samples will be collected for the analysis of clinical chemistry parameters.
Time Frame: Up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

15. Secondary Outcome: Number of Participants With Abnormal Ocular Findings on Ophthalmic Examination
Time Frame: Up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

16. Secondary Outcome: Plasma Concentrations of Belantamab Mafodotin (ADC)
Description: Blood samples will be collected for PK analysis of belantamab mafodotin.
Time Frame: Up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

17. Secondary Outcome: Plasma Concentrations of Monomethyl Auristatin-F With a Cysteine Linker (Cys-mcMMAF)
Description: Blood samples will be collected for PK analysis of belantamab mafodotin.
Time Frame: Up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

18. Secondary Outcome: Area Under Plasma Concentration-time Curve (AUC) From Time 0 to the Time of the Last Quantifiable Concentration (C(Tlast)) [AUC (0-last)] for Pomalidomide
Description: Blood samples will be collected for PK analysis of Pomalidomide in combination with belantamab mafodotin and dexamethasone
Time Frame: Up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

19. Secondary Outcome: Area Under Plasma Concentration-time Curve (AUC) From Time 0 to End of the Dosing Interval [AUC (0-tau)] for Pomalidomide
Description: as for outcome 18
Time Frame: Up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

20. Secondary Outcome: Maximum Concentration (Cmax) for Pomalidomide
Description: as for outcome 18
Time Frame: Up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

21. Secondary Outcome: Time of Cmax (Tmax) for Pomalidomide
Description: as for outcome 18
Time Frame: Up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

22. Secondary Outcome: Trough Concentration Prior to the Next Dose for Each Cycle (Ctrough) for Pomalidomide
Description: as for outcome 18
Time Frame: Up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

23. Secondary Outcome: Last Time Point Where the Concentration is Above the Limit of Quantification (Tlast) for Pomalidomide
Description: as for outcome 18
Time Frame: Up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

24. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADAs) Against Belantamab Mafodotin
Description: Serum samples will be collected for the analysis of the presence of ADAs using validated immunoassays. All samples will be tested in screening assay, and positive samples will be further characterized for antibody titers.
Time Frame: Up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

25. Secondary Outcome: Titers of ADAs Against Belantamab Mafodotin
Description: Serum samples will be collected for the analysis of the presence of ADAs using validated immunoassays. All samples will be further tested in screening assay, and positive samples will be further characterized for antibody titers.
Time Frame: Up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

26. Secondary Outcome: Number of Participants With Maximum Post-baseline Changes in Patient-reported Outcome Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) Scores for Each Item Attribute
Description: The PRO-CTCAE is a patient-reported outcome measure that was developed to evaluate symptomatic toxicities in patients in cancer clinical trials; it characterizes the frequency, severity, interference, and presence or absence of symptomatic toxicities. Responses ranges from 0 ("never," "none," "not at all," or "absent") to 4 ("almost constantly," "very severe," or "very much"), with a higher score indicating a higher frequency, severity, or interference of adverse events.
Time Frame: Up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

27. Secondary Outcome: Change From Baseline in Health Related Quality of Life (HRQoL) as Measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire 30-item Core Module (EORTC QLQ-C30)
Description: The EORTC QLQ-C30 includes 30-items with single and multi-item scales. These includes five functional scales (physical functioning [PF], role functioning [RF], cognitive functioning [CF], emotional functioning [EF] and social functioning [SF]), three symptom scales (fatigue, pain and nausea/vomiting [N/V]), a global health status (GHS)/ Quality-of-Life (QoL) scale, and six single items (constipation, diarrhoea, insomnia, dyspnoea, appetite loss [AL] and financial difficulties [FD]). Response options are 1 to 4. Scores are averaged and transformed to 0 to 100, a high score for functional scales/ GHS/QoL represent better functioning ability or health-related quality-of-life (HRQoL), whereas a high score for symptom scales/ single items represent significant symptomatology. Baseline is defined as latest pre-dose assessment (Day 1) with a non-missing value, including unscheduled visits. Change from Baseline is calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

28. Secondary Outcome: Change From Baseline in HRQoL as Measured by EORTC QLQ-20-item Multiple Myeloma Module (MY20)
Description: The EORTC Quality of Life Questionnaire 20-item Multiple Myeloma module (QLQMY20) is a supplement to the QLQ-C30 instrument used in participants with multiple myeloma. The individual component scores in the disease symptom domain are averaged and transformed linearly to a score ranging from 0 to 100. A high score for disease symptoms represents a high level of symptomatology or problems. A high score for Future Perspective and Body Image represents a high/healthy level of functioning. Baseline is defined as latest pre-dose assessment (Day 1) with a non-missing value, including unscheduled visits. Change from Baseline is calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

29. Secondary Outcome: Change From Baseline in HRQoL as Measured by EORTC Item Library 52 (IL52)
Description: The EORTC Quality of Life Questionnaire 20-item Multiple Myeloma module (QLQMY20) is a supplement to the QLQ-C30 instrument used in participants with multiple myeloma. For the EORTC IL52, disease symptoms domain of the QLQ-MY20 will be used for bone aches or pain, back pain, hip pain, arm or shoulder pain, chest pain, and pain increasing with activity. The individual component scores in the disease symptom domain are averaged and transformed linearly to a score ranging from 0 to 100. A high score for disease symptoms represents a high level of symptomatology or problems. Baseline is defined as latest pre-dose assessment (Day 1) with a non-missing value, including unscheduled visits. Change from Baseline is calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and up to approximately 407 weeks
Reporting Status: Not Posted, anticipated posting 2030-11

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected up to approximately 120 weeks. The results presented are until the primary completion date. Additional results will be provided within a year of study completion.
Description: Safety population included all randomized participants who received at least 1 dose of study intervention (any component).
Arm/Group | Belantamab Mafodotin+Pomalidomide+Dexamethasone | Bortezomib + Pomalidomide + Dexamethasone
All-Cause Mortality (participants affected / at risk) | 2/10 | 1/11
Serious Adverse Events (participants affected / at risk) | 5/10 | 4/11
Other Adverse Events (participants affected / at risk) | 10/10 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belantamab Mafodotin+Pomalidomide+Dexamethasone (N=10) | Bortezomib + Pomalidomide + Dexamethasone (N=11)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (2)
Oedema (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cytomegalovirus chorioretinitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Morganella infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (3) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belantamab Mafodotin+Pomalidomide+Dexamethasone (N=10) | Bortezomib + Pomalidomide + Dexamethasone (N=11)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (5)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (5) | 4 (11)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 3 (3) | 1 (1)
Dry eye (Eye disorders) | 2 (3) | 1 (2)
Eye discharge (Eye disorders) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 2 (4) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 4 (9) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (2) | 0 (0)
Vision blurred (Eye disorders) | 9 (17) | 1 (1)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (2)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (4)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 3 (4)
Localised oedema (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 3 (3) | 2 (2)
Oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 4 (4)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Hypogammaglobulinaemia (Immune system disorders) | 3 (4) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2)
Cystitis (Infections and infestations) | 1 (1) | 1 (6)
Dermatophytosis of nail (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (8)
Otitis externa (Infections and infestations) | 0 (0) | 1 (3)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Renal abscess (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (5) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (6)
Oral contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (8) | 2 (6)
Albumin urine present (Investigations) | 0 (0) | 1 (4)
Aspartate aminotransferase increased (Investigations) | 4 (6) | 1 (3)
Basophil count increased (Investigations) | 0 (0) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 3 (4) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (9)
Blood lactate dehydrogenase increased (Investigations) | 1 (2) | 0 (0)
Coagulation test abnormal (Investigations) | 1 (1) | 0 (0)
Cytomegalovirus test positive (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (2) | 3 (27)
Neutrophil count decreased (Investigations) | 3 (10) | 5 (45)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 3 (8) | 4 (12)
Weight decreased (Investigations) | 0 (0) | 1 (2)
White blood cell count decreased (Investigations) | 1 (2) | 4 (28)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (2)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Neurogenic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2025-01-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT06956170/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/70/NCT06956170/SAP_001.pdf